CLINICAL TRIAL: NCT06716931
Title: Investigating Benefits of A Physical Therapist (PT)-Guided Exercise Program in Myotonic Dystrophy Type 2 (DM2)
Brief Title: Investigating Exercise in Myotonic Dystrophy Type 2 (DM2)
Acronym: DM2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Paloma Gonzalez Perez, MD, PhD, Neurologist, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PGP-ZS
Record Dates: First submitted 2024-10-30; First posted 2024-12-04 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2024-11

CONDITIONS: Myotonic Dystrophy 2
Keywords: exercise; physical therapist; myotonic dystrophy type 2; electrical impedance myography
MeSH Terms: conditions — Myotonic Dystrophy; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Active Comparator): Exercise under the supervision of physical therapist in clinic during the first 3 months, then self-directed exercise routine for the last 3 months
  Interventions: Other: Exercise
- Group B (Active Comparator): Exercise under the supervision of physical therapist virtually during the first 3 months, then self-directed exercise routine for the last 3 months
  Interventions: Other: Exercise
- Group C (Active Comparator): Self-directed exercise routine for the first 3 months, then exercise routine under the supervision of physical therapist virtually during the last 3 months
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — A patient-friendly exercise routine has been designed for patients with myotonic dystrophy type 2. Benefits of this exercise regimen in different settings (at home versus clinic, self-directed versus physical therapist-directed) will be investigated.
  In person exercise supervised by physical therapist and then self-directed exercise in Group A
  Arms: Group A
Other: Exercise — Exercise virtually supervised by physical therapist and then self-directed for group B
  Arms: Group B
Other: Exercise — Self-directed and virtually supervised exercise by physical therapist for Group C
  Arms: Group C

SUMMARY:
An exercise regimen (PRIME: Proximal Resistance In-House Movement Exercise) has been designed for patients with myotonic dystrophy type 2 (DM2). The hypothesis is that this patient-friendly physical therapist (PT)-guided exercise program associates with improved functional capacity and muscle composition in DM2 in this two-period two-sequence cross-over study. Thus, participant will be randomized to one of the three possible groups. Participants in GROUP A will perform exercise routine in clinic under the direct supervision of a physical therapist twice a week for the first three months, then they will continue with same exercise routine at home for the last 3 months on their own. Participants in GROUP B will perform exercise routine virtually under the direct supervision of a physical therapist twice a week for the first three months, then they will continue with same exercise routine at home for the last 3 months on their own. Participants in GROUP C will perform exercise routine on their own during the first 3 months, then they will perform exercise routine virtually under the direct supervision of a physical therapist. Each group will include around 8 participants. Duration of the study is 6 months. In addition to exercise sessions, participants will have evaluation of their strength, motor function and muscle composition at three time points: initiation, 3 months and completion of the study at 6 months. Muscle composition will be assessed by electrical impedance myography which is a portable, non-invasive, painless and non-radiation tool that applies a weak high multifrequency electrical current to the examined muscle and allows to obtain information about its composition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with genetically confirmed myotonic dystrophy 2 (DM2) who are ≥18 and ≤ 70 years old.
* Patients are ambulatory without need of any assistance or device.
* Patients have a normal ECG within the 3 months prior to Screening visit (of note, patients with DM2 are recommended to have routine ECG as part of patient care. So, this ECG will be done as part of patient care).
* Body mass index (BMI) ≥20 and ≤30.

Exclusion Criteria:

* Subjects younger than 18 years old or older than 70 years old.
* Inability or unwillingness of the subject to give written informed consent.
* Subjects with pacemaker.
* Blood pressure <90/50 mmHg or >160 mmHg/90 mmHg at Screening visit
* Resting heart rate of <60 or >100 beats/minute at Screening visit.
* Any fall within the last six months.
* Any history of syncopal episodes or family history of sudden death.
* Patients who are pregnant or plan to become pregnant. A urine pregnancy test will be performed at visit 1 and 3 for women of childbearing age. If positive or if subject is planning to become pregnant, subject will be not eligible for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Manual Muscle Test (MMT) | From enrollment to the end of treatment at 6 months
  Score of manual muscle strength test scale. This is a strength exam at bedside of muscle groups
Six-minute walking test | From enrollment to the end of treatment at 6 months
  Distance in meters that subject can walk in six minutes

SECONDARY OUTCOMES:
Quantitative myometry | From enrollment to the end of treatment at 6 months
  Muscle dynamometry of different muscle groups measured in kilograms
Muscle resistance/reactance measures in ohms | From enrollment to the end of treatment at 6 months
  using electrical impedance myography, resistance and reactance measures in ohms will be obtained simultaneously from each examined muscle

OTHER OUTCOMES:
Time up to go | From enrollment to the end of treatment at 6 months
  Time in seconds from standing up, walk 3 meters, come back and sit again.
10 meter walk testing | From enrollment to the end of treatment at 6 months
  Time in seconds during a 10-meter walk.
Five times sit to stand | From enrollment to the end of treatment at 6 months
  Time in seconds to complete 5 times sit to stand.
Functional gait assessment (FGA) | From enrollment to the end of treatment at 6 months
  Assessment of balance using a scale (0-30) while walking and performing motor tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromuscular Diagnostic Center. Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided